CLINICAL TRIAL: NCT05669677
Title: Prospective Cohort Study to Determine the Response to COVID-19 Vaccination and Prevalence of COVID-19 in Subjects With Chronic Liver Disease
Brief Title: Study to Determine the Response to COVID-19 Vaccination and Prevalence of COVID-19 in Subjects With Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000118; 000118-DK
Record Dates: First submitted 2022-12-30; First posted 2023-01-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05-14

CONDITIONS: Chronic or Recovered Hepatitis B; Chronic or Recovered Hepatitis C; Chronic or Recovered Hepatitis D; NAFLD; NASH
Keywords: SARS-CoV-2; Liver Disease; Natural History
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard: Chronic liver disease

SUMMARY:
Background:

The COVID-19 global pandemic killed more than 6 million people worldwide. Several vaccines have been developed against the virus that causes this disease. These vaccines are effective at preventing severe symptoms and death from COVID-19. Some people with chronic liver disease, especially those with an advanced condition called cirrhosis, do not respond to many vaccines as well as healthy people do. The goal of this natural history study is to find out how well people with chronic liver disease respond to the COVID-19 vaccines.

Objective:

To learn how chronic liver disease affects the body s immune response to vaccination against COVID-19.

Eligibility:

People aged 18 years or older with chronic liver disease. They must also be enrolled in protocol 91-DK-0214 or 18-DK-0091.

Design:

Participants will have 3 visits, each spaced 6 months apart. Each visit will last 2 hours.

Participants will have their vital signs recorded. These include age, sex, race, height, and weight. They will give their medical history.

At each visit, participants will have blood drawn through a needle inserted into a vein in the arm. The sample drawn at each visit will be from 1 to 8 tablespoons.

At each visit, participants will fill out a questionnaire. They will answer questions about whether they have been vaccinated against COVID-19; whether they have had COVID-19; and whether they have been exposed to someone who had COVID-19. The questionnaire will take 10 to 15 minutes.

Researchers will also look at results of past blood tests from other research studies.

DETAILED DESCRIPTION:
Study Description:

The goals of this study are to assess the response to COVID vaccination in patients with chronic liver disease. Secondary goals are to evaluate the durability of antibody response against SARSCOV-2 and if SARS-COV-2 seropositivity is associated with reactivation or worsening of chronic hepatitis B.

Hypothesis:

Subjects with cirrhosis will have poorer response to COVID vaccination compared to subjects without cirrhosis and to healthy controls.

Objectives:

Primary Objective

To determine the response to SARS-COV-2 vaccination among patients with chronic liver disease stratified by severity (cirrhosis vs no cirrhosis) and compare to healthy controls

Secondary Objectives

* To determine the durability of antibody against SARS-COV-2 among patients with chronic liver disease
* To determine if SARS-COV-2 seropositivity is associated with reactivation or worsening of chronic hepatitis B

Tertiary Objective

* To determine how SARS-COV-2 affects the pre-existing HBV, HCV, HDV-specific immune response of subjects with liver disease via T cell receptor cross-reactivity or cytokine-mediated bystander cell activation
* To determine whether T and B responses to SARS-COV-2 infection or SARS-COV-2 vaccination differ in subjects with and without chronic liver disease and with and without liver cirrhosis.
* To determine whether antibody and T and B cell responses against polyethylene glycol (PEG) increase over time and affect the response to the covid vaccine.

Endpoints:

Primary Endpoints

The proportion of patients with >100 BAU/mL SARS-COV2 antibody levels one year after Covid-19 vaccination

Secondary Endpoints

* Changes in levels of SARS- COV-2 antibody over time among patients with chronic liver disease stratified by severity (cirrhosis vs no cirrhosis) compared to healthy controls
* Assess prevalence of HBV reactivation, defined as reappearance of HBsAg in serum and/or reappearance or increase in HBV DNA by 1 log10 IU/mL in serum in patients with and without prior Covid-19

Tertiary Endpoint

* Comparison of HBV, HCV and HDV-specific immune responses before and after SARS-COV-2 infection in patients who experienced SARS-COV-2 between study time points or using as pre-infection time point PBMC stored prior to November 2019 (first global report of SARS-COV-2)
* Comparison of T and B responses to SARS-COV-2 infection or SARS-COV-2 vaccines in subjects with and without chronic liver disease and with and without liver cirrhosis, and evaluation of durability of responses in subsequent study visit.
* Assessment of anti-PEG IgM and IgG levels and T and B responses against PEG.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to participate in this study, an individual must meet all of the following criteria:

1. Male or females >= 18 years of age
2. Evidence of chronic liver disease within the last 12 months.

   a. Patients with chronic hepatitis B who became negative for HBsAg will be eligible because they may reactivate following SARS-COV-2 exposure.
3. Enrolled in protocol 91-DK-0214 or 18-DK-0091

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of only resolved chronic Hepatitis C (anti-HCV positive, HCV RNA negative) with no evidence of any other chronic liver disease, unless cirrhotic or unless prior cryopreserved peripheral blood mononuclear cells (PBMC) available.
2. Inability to provide informed consent
3. Patients with primary immunodeficiency disorders
4. Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects greater than or equal to 18 years of age will be recruited from study 91-DK-0214: with chronic liver disease or recovery of chronic liver disease followed at the Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARSCOV-2 in subjects with chronic liver disease | ongoing
  To determine the response to SARS-COV-2 vaccination among patients with chronic liver disease stratified by severity (cirrhosis vs no cirrhosis) and compare to healthy controls

SECONDARY OUTCOMES:
To determine the durability of antibody against SARS-COV-2 among patients with chronic liver disease. | ongoing
  Changes in quantitative levels of SARS-COV-2 antibody over time
To determine if SARS-COV-2 seropositivity is associated with reactivation or worsening of chronic hepatitis B. | ongoing
  Prevalence of HBV re-activation among patients with and without exposure to SARS-COV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Since the clinical significance of COVID antibody test results is unclear, we do not plan to inform subjects of these results. Should participants be interested in their current COVID status, we will refer them to testing clinics or to their primary provider for PCR testing.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000118-DK.html